CLINICAL TRIAL: NCT01585948
Title: The Role of Newer and Traditional Risk Factors in the Development, Extent and Manifestation of Coronary Artery Disease
Brief Title: Study of the Effect of Diabetes on the Incidence and the Extent of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: University of Ioannina (Other)
Collaborators: University Hospital, Ioannina (Other); Catheterization Laboratory of 1st IKA Hospital, Athens (Unknown)
Responsible Party: Principal Investigator, MICHALIS LAMPROS, Professor of Cardiology, Medical School, University of Ioannina, University of Ioannina
Other Study IDs: UOICAD2010
Record Dates: First submitted 2011-08-16; First posted 2012-04-26 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Patients Undergoing Coronary Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Includes retaining blood samples for DNA analyses and biochemical markers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Diabetes Mellitus: All patients undergoing coronary angiography who are diabetics.
- No diabetes mellitus: All patients undergoing coronary angiography that are non-diabetics.
- Coronary angiography patients: Diabetics and non-diabetics with or without known CV disease who are admitted in the Department of Cardiology in the University Hospital of Ioannina and the Catheterization Laboratory of 1st IKA Hospital in Athens and undergo coronary angiography for clinical purposes will be studied. The study will include subjects who 1) have suspected CAD and undergo a scheduled diagnostic angiogram for clinical reasons, and 2) are hospitalized because of an acute coronary syndrome and thus undergo diagnostic angiography (with or without previous history of CAD).

SUMMARY:
In the present study the investigators will measure the extent of coronary artery disease via coronary angiography and the correlating risk factors.

DETAILED DESCRIPTION:
In the present study the investigators will examine the risk factors determining the development, extent and the manifestation of coronary artery disease. The study will recruit patients undergoing coronary angiography for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* Any subject eligible for coronary angiography with or without known CV disease for clinical reasons.

Exclusion Criteria:

* Patients revascularized in the past, with either coronary artery bypass grafting or percutaneous coronary intervention, will be excluded from the study since it is not possible to describe the extent of CAD in these patients.
* Moderate or severe aortic stenosis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetics and non-diabetics who are admitted in the Cardiology Department in the University Hospital of Ioannina and undergo coronary angiography for clinical purposes will be studied. The study will include subjects who have suspected stable CAD or an acute coronary syndrome and undergo a diagnostic angiography. Patients revascularized in the past (either coronary artery bypass grafting or percutaneous coronary intervention) will be excluded from the study since it is not possible to describe the extent of CAD in these patients.
  We plan to recruit about 1,000 patients in about 2 years in order for valid conclusions to be drawn from association analysis between CV risk factors, gene polymorphisms and the presence and extent of CAD.
Sampling Method: Probability Sample
Enrollment: 1104 (Actual)
Dates: Start 2009-11; Primary Completion 2013-05 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
The incidence and extent of coronary artery disease between diabetics and non-diabetic patients. | Up to four years on average.
  We will investigate the incidence, extent and clinical manifestation of coronary artery disease in diabetics and non-diabetics undergoing coronary angiography for clinical reasons.

SECONDARY OUTCOMES:
The incidence and extent of coronary artery disease via coronary angiography scores and related biochemical and demographical risk factors. | Up to 4 years on average.
  To associate the incidence, extent and clinical manifestation of coronary artery disease with classic demographic risk factors (such as smoking, alcohol consumption, physical exercise, arterial hypertension, family history of diabetes mellitus or coronary artery disease) and common biochemical risk factors (such as fasting glucose levels, urea, creatinine, HbA1c%, uric acid, total cholesterol, HDL, LDL, triglycerides, VLDL, glomerular filtration rate - GFR).
The incidence, extent and clinical manifestation of coronary artery disease and the circulating levels of hs-CRP, adipokines and RAGEs. | Up to 4 years on average.
  To associate the incidence, extent and clinical manifestation of coronary artery disease with systemic inflammatory status assessed by hs-CRP levels, circulating adipokines (adiponectin, resistin) and the receptors of advanced glycation end products (sRAGE and esRAGE).
TCF7L2 gene polymorphims and the incidence and extent of coronary artery disease. | Within a maximum period of 4 years.
  To associate the incidence, extent and clinical manifestation of coronary artery disease with the rs7903146 single nucleotide polymorphism of TCF7L2 gene, that has been strongly associated with diabetes mellitus development.

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Naka, As Professor, Principal Investigator — University of Ioannina
Locations (1):
- 2nd Department of Cardiology, University Hospital of Ioannina, Ioannina, Greece